CLINICAL TRIAL: NCT06315751
Title: A Double-blind, Placebo-controlled, Phase 2b, Multi-center, Twelve-week Prospective Study to Evaluate the Efficacy and Safety of Gemlapodect in Adult and Adolescent Patients With Tourette Syndrome
Brief Title: Efficacy and Safety of Gemlapodect (NOE-105) in Adults and Adolescents With Tourette Syndrome
Acronym: ALLEVIA2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Noema Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NOE-TTS-201
Record Dates: First submitted 2023-12-06; First posted 2024-03-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-05

CONDITIONS: Tourette Syndrome
Keywords: NOE-105
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gemlapodect (Experimental): Escalating doses of NOE-105 capsules
  Interventions: Drug: Gemlapodect
- Placebo (Placebo Comparator): Escalating doses of matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gemlapodect — Gemlapodect is an investigational selective PDE10A inhibitor with a potential therapeutic effect for the treatment of tics associated with TS. Administered in the form of oral capsules.
  Other Names: NOE-105
  Arms: Gemlapodect
Drug: Placebo — Administered in the form of oral capsules with inert ingredients.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy and safety of gemlapodect (NOE-105) on reducing tics associated with Tourette Syndrome (TS) in adults with TS. Adolescents will be enrolled after a sentinel cohort of adults is complete.

DETAILED DESCRIPTION:
Gemlapodect is an investigational selective PDE10A inhibitor with a potential therapeutic effect for the treatment of tics associated with Tourette Syndrome (TS). This is a multi-center, double-blind, parallel-arm, placebo-controlled study in patients with TS. Following screening to confirm eligibility and to wash-out previous TS medication during a 14-day placebo run-in, patients will be randomized 1:1 on Day 1 to receive gemlapodect or placebo once daily for 12 weeks. See https://allevia2study.com

ELIGIBILITY:
Inclusion Criteria:

1. Initially, patients aged 18 years onwards, at the time of signing the ICF form. Adolescents aged 12 years and older at the time of signing the ICF/informed assent form will be eligible for inclusion after completion of a sentinel cohort of adults.
2. Moderate to severe Tourette Syndrome as defined by DSM-5 diagnostic criteria and TS-CGI-S ≥ 4.
3. Treatment naive or previously treated patients in need of treatment alternative as per investigators judgement.
4. Patients must discontinue all medications used to treat TS for at least 14 days prior to randomization. Other psychotropic drugs, including stimulants, will be allowed provided they have been stable for at least 30 days prior to randomization and are expected to remain stable for the duration of the study.
5. BMI within the range 18 to 35 kg/m2 (inclusive).
6. Women of childbearing potential should only be included after a confirmed menstrual period and a negative highly sensitive urine or serum pregnancy test. Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
7. Capable of giving signed informed consent or consent from their legal representative.
8. Fluency in the language of the investigator, study staff, and the ICF/informed assent form when applicable.

Exclusion Criteria:

1. Any medical condition which, in the opinion of the investigator, could interfere with study procedures including but not limited to functional tic-like disorder, secondary tic symptoms accompanied by late-onset tics, Huntington's chorea, malignant TS, neuroacanthocytosis, autism, and history of known intellectual disability that would affect patient's ability to comply with study procedures.
2. Current active diagnosis of severe anxiety, bipolar disorder, schizophrenia, major depressive disorder (MDD,), or Parkinson's disease. Patients with a history of MDD on selective serotonin reuptake inhibitors treatment stable for at least a month may participate in the study.
3. A history of severe traumatic brain injury or stroke.
4. Any unstable medical conditions, severe symptoms, or clinically significant abnormalities on screening test/examinations, including uncontrolled seizure disorders, which, in the investigator's judgment, will put them at a risk of major AE during this trial, or will interfere with safety and efficacy assessments.
5. Are undergoing active CBT (including but not limited to comprehensive behavioral intervention for tics, exposure and response prevention, relaxation training) during the last 28 days before the planned date of randomization and until the end of the trial. Patients willing to discontinue their CBT over this period are eligible to enroll in the study.
6. Known DSM-5 diagnosis of substance abuse or dependence.
7. Active suicidal ideation or behavior.
8. Use of prescribed or recreational cannabinoids during the study are prohibited. Prescribed cannabinoids include Epidiolex® (cannabidiol), Marinol® /Syndros® (dronabinol), and Cesamet® (nabilone). These medications will be discontinued during the Screening period. Study participants prescribed cannabinoids for seizure disorders are not eligible for study participation. Recreational cannabinoids, regardless of their form of intake, which include tetrahydrocannabinol and/or cannabidiol, are prohibited.
9. Strong inhibitors and inducers of CYP3A4 are prohibited during the study.
10. Neurostimulation/deep brain stimulation for TS.
11. Participation in another clinical study with a study intervention administered in the last 30 days.
12. Patients with a known hypersensitivity to gemlapodect or any of the excipients of the product
13. Positive urine drug screen for cannabis, cocaine, or nonprescribed opiates.
14. The person is an employee or family member of an employee of the Sponsor, Investigator, or study site personnel.
15. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
16. Previous randomization in the present study.
17. The person is currently committed to an institution by virtue of an order issued either by the judicial or the administrative authorities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in tic severity score on the Revised Yale Global Tic Scoring Scale (YGTSS-R) | 85 days
  YGTSS-R is a clinician rated score that evaluates number, frequency, intensity, complexity and interference of motor and phonic tics with a total score ranging from 0 to 50, with 50 being the most severe and 0 being no tics. Change in YGTSS-R total tic scores from baseline (randomization) to D85 for gemlapodect as compared to placebo.
  The primary estimand is the difference in means between gemlapodect and placebo for the change in the TTS of the YGTSS-R from baseline (randomization) to D85, in the target patient population of adult and adolescent patients with TS, regardless of whether or not dose reduction, suspension, or treatment discontinuation occurred due to events attributable to treatment, and regardless of change in background medication (dose and product) while under treatment, but in the absence of any new treatment started after discontinuation of investigational intervention

SECONDARY OUTCOMES:
Impact on patient functioning | 85 days
  Change in Sheehan Disability Scale from baseline (randomization) to D85 for gemlapodect as compared to placebo
Change in PUTS | 85 days
  Change in premonitory urge for tics scale from baseline (randomization) to D85 for gemlapodect as compared to placebo
Safety and Tolerability of gemlapodect | 85 days
  The Incidence and severity of adverse events, including serious adverse events and adverse events of special interest
Assessment of suicidality and suicidal ideation | 85 days
  Change in Columbia Suicide Severity Rating Scale (C-SSRS) subscale from baseline(randomization) to D85 for gemlapodect as compared to placebo. The C-SSRS supports suicide risk assessment through a series of simple, plain-language questions to assesses suicidal ideation and suicidal behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, MD, Study Director — Noema Pharma AG
Locations (46):
- United States (31):
  - Noema TTS-201 Site #81, Sun City, Arizona
  - Noema TTS-201 Site #95, Bellflower, California
  - Noema TTS-201 Site #75, Glendale, California
  - Noema TTS-201 Site #59, San Rafael, California
  - Noema TTS-201 Site #21, Walnut Creek, California
  - Noema TTS-201 Site #54, Gulf Breeze, Florida
  - Noema TTS-201 Site #05, Hialeah, Florida
  - Noema TTS-201 Site #97, Jensen Beach, Florida
  - Noema TTS-201 Site #71, Largo, Florida
  - Noema TTS-201 Site #44, Maitland, Florida
  - Noema TTS-201 Site # 74, Miami, Florida
  - Noema TTS-201 Site #56, Miami Lakes, Florida
  - Noema TTS-201 Site #61, Orlando, Florida
  - Noema TTS-201 Site #79, Atlanta, Georgia
  - Noema TTS-201 Site #87, Peachtree Corners, Georgia
  - Noema TTS-201 Site #55, Boston, Massachusetts
  - Noema TTS-201 Site #51, Ann Arbor, Michigan
  - Noema TTS-201 Site #96, Saint Charles, Missouri
  - Noema TTS-201 Site #93, Lincoln, Nebraska
  - NOema TTS-201 Site #19, New York, New York
  - Noema TTS-201 Site #03, Stony Brook, New York
  - Noema TTS-201 Site #57, Charlotte, North Carolina
  - Noema TTS-201 Site #58, Middleburg Heights, Ohio
  - Noema TTS-201 Site #73, North Charleston, South Carolina
  - Noema TTS-201 Site #98, Nashville, Tennessee
  - Noema TTS-201 Site #42, Dallas, Texas
  - Noema TTS-201 Site #22, Fort Worth, Texas
  - Noema TTS-201 Site #94, San Antonio, Texas
  - Noema TTS-201 Site #45, Orem, Utah
  - Noema TTS-201 Site #18, Petersburg, Virginia
  - Noema TTS-201 Site #50, Bellevue, Washington
- Noema TTS-201 Site #06, Ghent, Belgium
- France (2):
  - Noema TTS-201 #07, Bron
  - Noema TTS-201 Site #08, Poitiers
- Germany (3):
  - Noema TTS-201 Site #35, Düsseldorf
  - Noema TTS-201 Site #09, Hanover
  - NOE-TTS-201 Site #25, Munich
- Noema TTS-201 Site #30, Budapest, Hungary
- Poland (2):
  - Noema TTS-201 Site #13, Katowice
  - Noema TTS-201 Site #14, Katowice
- Spain (6):
  - Noema TTS-201 Site #26, Barcelona
  - Noema TTS-201 Site #15, Burgos
  - Noema TTS-201 Site #27, Madrid
  - Noema TTS-201 Site #17, Oviedo
  - Noema TTS-201 Site #16, Sant Cugat del Vallès
  - NOE-TTS-201 Site #28, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://allevia2study.com/